CLINICAL TRIAL: NCT04521894
Title: Diagnostic Performance of 18F-prostate-specific Membrane Antigen-1007 PET/CT in the Detection of Prostate Cancer
Brief Title: The Application Value of 18F-prostate-specific Membrane Antigen PET/CT in Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019LunShenYiZiDiJ1Hao; XJTU1AF-CRF-2020-008 (Other: the First Affiliated Hospital of Xian Jiaotong University)
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate-specific antigen; PET/CT; PSMA; Gleason Score
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron-Emission Tomography; Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Primary PCa without metastases Group: Participants who are suspected of prostate cancer due to elevated PSA or clinical symptoms but have not received any treatment and eventually confirmed prostate cancer after surgery or biopsies.
  Interventions: Device: Positron emission tomography/computerized tomography (PET/CT)
- Primary PCa with metastases Group: Participants who are suspected of prostate cancer due to elevated PSA or clinical symptoms but have not received any treatment and eventually confirmed prostate cancer after surgery or biopsies. And the 18F-PSMA-PET/CT scan confirmed metastases.
  Interventions: Device: Positron emission tomography/computerized tomography (PET/CT)
- Oligometastatic PCa group: "Oligometastatic"is a subgroup of metastatic patients with a limited number of secondary lesions (threshold ranging from 3 to 5) in one or few organs.
  Interventions: Device: Positron emission tomography/computerized tomography (PET/CT)
- Biochemical recurrence Group: Proven biochemical recurrence after radical therapy (PSA >0.2 ng/mL after radical prostatectomy, PSA ≥2 ng/mL above the nadir after external-beam radiotherapy) or persisting PSA after radical treatment with rising PSA values.
  Interventions: Device: Positron emission tomography/computerized tomography (PET/CT)
- Control Group: Prostate cancer benign prostatic hypertrophy or normal prostate.
  Interventions: Device: Positron emission tomography/computerized tomography (PET/CT)

INTERVENTIONS:
Device: Positron emission tomography/computerized tomography (PET/CT) — 1. Genetic factors and age:
     Epidemiological studies have shown that if an immediate family member (brother or father) suffers from prostate cancer, the risk of prostate cancer will be more than doubled. Age is a relatively strong risk factor for PCa.
  2. Prostatitis: Prostatitis is related to PCa. Cancer is usually found in the tissues where inflammation is found.
  3. Obesity: Research has found that obese patients have a low grade of PCa, but their risk of developing aggressive cancer is higher.
  4. Infection:
  5. Exercise: Most studies have found that exercise does not reduce the risk of prostate cancer, but some studies have shown that.
  6. Daily diet: The corrective mechanism of diet in PCa is not very clear.
  7. Drinking history:

SUMMARY:
Prostate cancer (PCa) is the most common type of malignant tumor and the third leading cause of cancer-associated mortality among men worldwide. The biological behaviors of PCa at different degrees of malignancy also largely differ, directly impacting disease outcomes and responses to treatment. Therefore, accurate risk stratification of PCa before treatment and the development of an individualized treatment regimen, play a vital role to improve the clinical outcome of patients. However, overdiagnosis and unnecessary biopsies, which are invasive examinations associated with higher costs and adverse effects. When the PSA is less than 20ng/mL, less than 1% of PCa patients have a positive bone scan, and routine bone scans are not recommended for asymptomatic or low-risk PCa patients. Interestingly, due to the variations among evaluators that often occur when defining the T stage, biopsies operate inaccuracy, also low-PSA level can also occur metastasis, there is a need for an objective and accurate imaging biomarker for the diagnosis of different grade PCa.

Prostate-specific membrane antigen (PSMA) is a type II transmembrane protein, which has higher expression in cancerous prostate cells than in normal prostate cells. Meanwhile, its expression level is positively correlated with the degree of malignancy, the tendency of metastasis, and the risk of early recurrence. In recent years, 18F-PSMA positron emission tomography/computerized tomography (PSMA PET/CT) has earned widespread attention as a novel imaging modality based on molecular-level analysis, rather than morphological or physiological analysis, to assist in PCa diagnosis and tumor burden evaluation.

Currently, Maximum Standardized Uptake Value (SUVmax) is the most commonly used semi-quantitative parameter in PET/CT, which is used to assess tumor burden of PCa, and thus can be used as an imaging biomarker to assess the degree of malignancy of prostate cancers. However, prior studies mainly focused on the correlation between patients' biochemical recurrence lesions and the PSA levels and Gleason score. There is a lack of research to explore the correlation among primary PCa burden, PSA levels, and the degree of prostate cancer malignancy. The aim of this project is to use 18F-PSMA PET/CT SUVmax to analyze the correlation among primary PCa imaging, and clinical indicators, and to evaluate the predictive value for PCa risk stratification, metastasis risk, and biochemical recurrence.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the highest malignant male tumor and one of the leading causes of mortality among men worldwide. The biological behaviors of PCa malignancy are largely heterogeneous, directly impacting prognostic grouping and treatment options. In addition, assessments of the distant metastatic status for PCa patients have recently received increasing attention due to the heightening mortality rate. Therefore, the precise systemic staging of primary PCa risk stratification before treatment plays a crucial role in designing the management strategy for the individualized treatment option. According to both American Urological Association (AUA) and the European Association of Urology (EAU) guidelines, patients with total prostate-specific antigen (tPSA) > 20 ng/mL and/or Gleason Score ≥ 8 are high-risk, the probability of distant metastasis and mortality will increase significantly and may not suitable for active surveillance programs, radical prostatectomy or radiotherapy treatment. However, tPSA is organ-specific but not tumor-specific, the biological behaviors of prostate malignancy are largely heterogeneous, and the specificity of the ability of tPSA to reflect distant metastasis remains debatable. Using tPSA as the only indicator for risk stratification discrimination and distant metastases prediction may causing in large numbers of unnecessary prostate biopsies. Also, elderly patients with severe comorbidities or undergoing anticoagulation therapy may not be the optimal candidates for biopsies and may cause adverse effects and higher costs. In these cases, it is urgent to find objective and accurate imaging biomarkers for risk stratification classification with a noninvasive approach based on imaging analysis.

The prostate-specific membrane antigen (PSMA) is a type II transmembrane glycoprotein that is primarily expressed in prostatic tissues, and its expression is correlated with the degree of malignancy and further increases in metastatic. The ability of PSMA to easily penetrate tissues and diffuse with solid tumor lesions can reflect the statuses of metastasis. Prior studies show that PSMA PET/CT is superior to conventional imaging methods for lymph node metastatic detection and that the pre-treatment tPSA level and Gleason Score are associated with the PSMA uptake in primary PCa. Furthermore, the Maximum Standardized Uptake Value (SUVmax) is the most commonly used semi-quantitative parameter in PET/CT and prior studies have already been used to assess the degree of malignancy of PCa and predict extended pelvic lymph node metastases in intermediate to high-risk PCa patients by 68Ga-PSMA-11 or 68Ga-PSMA-617. 18F-PSMA-1007 is advantaged by its higher spatial resolution images and non-urinary excretion that reduces urinary clearance, this approach bears a great potential to facilitate the detection of primary PCa and metastatic lesions. However, to our knowledge, no prior studies have employed 18F-PSMA-1007 PET/CT to evaluate the diagnostic performance in risk stratification and distant metastases prediction in primary PCa.

The present study aims to retrospective investigated the role of 18F-PSMA-1007 PET/CT semi-quantitative parameters correlation among newly diagnosed PCa imaging, tPSA levels and Gleason Score, and to evaluate the prediction performance of 18F-PSMA-1007 PET/CT and clinicopathologic characteristics on PCa risk stratification and distant metastatic prediction.

ELIGIBILITY:
Inclusion Criteria:

* 1 age between 40 and 100 years old
* 2 PSA >0.4 ng/mL for primary PCa with biopsy proven or RP diagnosis of prostate cancer
* 3 PSA >0.2 ng/mL after RP, PSA ≥2 ng/mL above the nadir after EBRT) or persisting PSA after radical treatment with rising PSA values
* 4 complete clinical, pathological, imaging and biochemical information

Exclusion Criteria:

* 1 lack of histological examinationproven diagnosis of PCa
* 2 18F-PSMA PET/CT being performed after pharmacotherapy since PSMA-targeted imaging can be disturbed by previous therapie

Ages: 40 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prostate cancer, benign prostatic hyperplasia, and healthy volunteers who are pathologically confirmed in the First Affiliated Hospital of Xi'an Jiaotong University due to elevated PSA levels or clinical symptoms will include in this study, with complete clinical and pathological data, and complete PET/CT scan before receiving treatment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-22 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax | From the time the participants first go to the hospital without treatment and through study completion, an average of 1 year. If the patient undergoes radical prostatectomy, an additional scan will be added within 1 month after surgery
  Maximum Standardized Uptake Value (SUVmax) is the most commonly used semi-quantitative parameter in PET/CT, which is used to assess tumor burden of PCa.
PSA | Through study completion, an average of 6 months
  Prostate-specific antigen, or PSA, is a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis. The results are usually reported as nanograms of PSA per milliliter (ng/mL) of blood.
Gleason Score | Baseline of the study by prostate cancer biopsies or after radical prostatectomy, and when there is a biochemical recurrence, an additional biopsies the prostate bed within 1 month.
  The cells are graded on a scale of 1 to 5. Grade 1 cells resemble normal prostate tissue. Cells closest to 5 are considered "high-grade" and have mutated so much that they barely resemble normal cells.

SECONDARY OUTCOMES:
BMI | Through study completion, an average of 6 months.
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness. BMI can be used to screen for weight categories that may lead to health problems but it is not diagnostic of the body fatness or health of an individual.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyi Duan, Ph.D., Study Chair — First Affiliate Hospital of Xi'an Jiaotong University
Locations (1):
- First Affiliate Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Luo L, Zheng A, Chang R, Li Y, Gao J, Wang Z, Duan X. Evaluating the value of 18F-PSMA-1007 PET/CT in the detection and identification of prostate cancer using histopathology as the standard. Cancer Imaging. 2023 Nov 3;23(1):108. doi: 10.1186/s40644-023-00627-x. PMID 37924154